CLINICAL TRIAL: NCT06458192
Title: Adaptive Messaging to Support Depression Self-Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rachel Kornfield, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00214828
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adaptive Messaging Intervention (Experimental): The intervention involves 8 weeks of daily text messaging. Messages will arrive throughout the day via SMS to prompt learning and applying cognitive and behavioral self-management strategies, representing a variety of self-management strategies and message tones. The intervention will apply reinforcement learning to select daily messaging styles to maximize user engagement.
  Interventions: Behavioral: Adaptive Messaging Intervention
- Non-Adaptive Messaging Intervention (Experimental): The intervention involves 8 weeks of daily text messaging. Messages will arrive throughout the day via SMS to prompt learning and applying cognitive and behavioral self-management strategies, representing a variety of self-management strategies and message tones. Daily messaging styles will be randomly selected.
  Interventions: Behavioral: Non-Adaptive Messaging Intervention
- Psychoeducation-only control (Active Comparator): The 8-week intervention involves receiving several text messages per week that include weblinks to access psychoeducation information about cognitive and behavioral self-management strategies.
  Interventions: Behavioral: Psychoeducation-Only Control

INTERVENTIONS:
Behavioral: Adaptive Messaging Intervention — The intervention delivers 8 weeks of daily text messaging. Messages will arrive throughout the day via SMS to prompt learning and applying cognitive and behavioral self-management strategies, representing a variety of self-management strategies and message tones. The intervention will apply reinforcement learning to select daily messaging styles to maximize user engagement.
  Other Names: Small Steps SMS
  Arms: Adaptive Messaging Intervention
Behavioral: Non-Adaptive Messaging Intervention — The intervention involves 8 weeks of daily text messaging. Messages will arrive throughout the day via SMS to prompt learning and applying cognitive and behavioral self-management strategies, representing a variety of self-management strategies and message tones. Daily messaging styles will be randomly selected.
  Other Names: Small Steps SMS
  Arms: Non-Adaptive Messaging Intervention
Behavioral: Psychoeducation-Only Control — An active control which will deliver psychoeducational content via clickable URLs over 8 weeks.
  Arms: Psychoeducation-only control

SUMMARY:
This is a pilot randomized controlled trial of an adaptive 8-week text messaging intervention for depression self-management. Among 100 individuals with elevated depression symptoms, the investigators will compare the effects of 8 weeks of the adaptive text messaging intervention (n=40) to 8 weeks of a non-adaptive text messaging intervention (n=40), and 8 weeks of a psychoeducation-only intervention (n=20). The investigators will include a 6-month post-treatment follow-up to verify that treatment gains are maintained.

Both messaging arms will receive 8 weeks of daily text messaging. Messages will prompt learning and applying cognitive and behavioral self-management strategies. Whereas the non-adaptive messaging system will randomly select daily messaging styles (representing a variety of self-management strategies and message tones), the adaptive messaging system will apply reinforcement learning to select daily messaging styles to maximize user engagement. Text messages will also be used to solicit feedback such as message ratings to inform the reinforcement learning algorithm (if applicable). The psychoeducation control group will receive a few brief text messages per week providing weblinks to access psychoeducation information.

The investigators will recruit participants through digital methods (e.g., advertising on social media platforms like Facebook and Instagram).

Administration of study measures will occur at baseline, weeks 4 and 8, and 3-month and 6-month follow-up. The primary outcomes is depression symptom severity (PHQ-9). Secondary outcomes are: anxiety severity (GAD-7) and suicidality (DSI-SS). Using an Intention to Treat paradigm, the investigators will test our hypothesis that:

H1: Relative to the psychoeducation-only control, messaging interventions will reduce depression (H1a) and anxiety and suicidal ideation (H1b).

H2: Relative to non-adaptive messaging, adaptive messaging will reduce depression (H1a) and anxiety and suicidality (H2b).

H3: Adaptive messaging will reduce depression relative to non-adaptive messaging by producing greater objective and subjective engagement.

DETAILED DESCRIPTION:
The primary goal of this prospective randomized controlled trial is to pilot all trial procedures for a larger, fully-powered trail. The investigators will enroll 100 participants out of consideration for feasibility.

Among individuals with elevated depression symptoms, the investigators will compare the effects of 8 weeks of an adaptive text messaging intervention (n=40), 8 weeks of a non-adaptive text messaging intervention (n=40), and a psychoeducation-only control group (n=20). The investigators will include a 6-month post-treatment follow-up to verify that treatment gains are maintained.

The study will enroll individuals who have at least moderate symptoms of depression as indicated by Patient Health Questionnaire-9 (PHQ-9) scores greater than or equal to 10.

The investigators will recruit participants through digital methods (e.g., advertising on social media platforms like Facebook and Instagram). Recruitment advertisements will direct potential participants to a centralized recruitment website that provides additional information about the IRB-approved protocol. Participants will represent likely users of a mobile-based depression intervention. They will also reflect the racial and ethnic diversity of the United States. Interested individuals will confirm eligibility by completing an online screening survey. Participants will self-report their specific recruitment source as part of this survey and will provide contact information. If eligible participants confirm interest, study staff will obtain informed consent.

Computer-generated randomization will be created prior to the start of the study to avoid allocation bias. Random block sizes of 5 and 10 will be allocated in a 2:2:1 ratio to adaptive messaging, non-adaptive messaging, and the psychoeducation-only control group.

Both messaging arms will receive 8 weeks of daily text messaging. Messages will prompt learning and applying cognitive and behavioral self-management strategies. Whereas the non-adaptive messaging system will randomly select daily messaging styles (representing a variety of self-management strategies and message tones), the adaptive messaging system will apply reinforcement learning to select daily messaging styles to maximize user engagement. Text messages will also be used to solicit feedback such as message ratings to inform the reinforcement learning algorithm (if applicable). The psychoeducation control group will receive a few brief text messages per week providing weblinks to access psychoeducation information.

Administration of study measures will occur as part of the research protocol via REDCap online at baseline, weeks 4 and 8, and 3-month and 6-month follow-up. The primary outcomes is depression symptom severity (PHQ-9). Secondary outcomes are: anxiety severity (GAD-7) and suicidality (DSI-SS). The investigators will additionally assess subjective and objective engagement with the intervention (messaging arms only).

The investigators will collect qualitative data with a subset of 10 participants in each messaging arm via user interviews.

Using an Intention to Treat paradigm, the investigators will use longitudinal linear mixed-effects models to test our hypothesis that:

H1: Relative to the psychoeducation-only control, messaging interventions will reduce depression (H1a) and anxiety and suicidal ideation (H1b).

H2: Relative to non-adaptive messaging, adaptive messaging will reduce depression (H1a) and anxiety and suicidality (H2b).

H3: Adaptive messaging will reduce depression relative to non-adaptive messaging by producing greater objective and subjective engagement.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* At least moderate depressive symptom severity (a score of 10 or higher on the PHQ-8)
* Has a smartphone
* Is able to speak and read English
* US citizen or resident

Exclusion Criteria:

* Reports diagnosis with a severe mental health problem (e.g., psychotic, bipolar) for which participation in this trial is inappropriate
* High suicide risk (has ideation, plan, and intent)
* Is currently receiving psychotherapy or intends to commence it in the next 8 weeks
* Psychiatric medication dose change in the past 4 weeks, or has plans to change the dose of a psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Assessments will be completed at baseline, week 4, week 8, week 20 (3 month follow-up) and week 32 (6 month follow-up).
  PHQ-9 is a 9-item questionnaire which produces a single score between 0 and 27, with higher scores indicating greater depression symptom severity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | Assessments will be completed at baseline, week 4, week 8, week 20 (3 month follow-up) and week 32 (6 month follow-up).
  GAD-7 is a 7-item questionnaire screening for symptoms of generalized anxiety disorder.
Depressive Symptom Index-Suicidality Subscale (DSI-SS) | Assessments will be completed at baseline, week 4, week 8, week 20 (3 month follow-up) and week 32 (6 month follow-up).
  DSI-SS is a brief (4-item) screening tool for suicidal symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this project may be shared with other investigators who provide a proposal with a strong research question and appropriate rationale and analytic plan. In such a case, data would be de-identified as per HIPAA regulations to protect the confidentiality of participants, and the investigators would work closely together to ensure high quality output and meet all compliance regulations of participating institutions.